CLINICAL TRIAL: NCT06467734
Title: Prospective Cohort Study of Synovial Biomarkers in the Diagnosis and Prediction of Periprosthetic Joint Infection
Acronym: Yes
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Long Hua, Doctor, First Affiliated Hospital of Xinjiang Medical University
Other Study IDs: XJ202405-02
Record Dates: First submitted 2024-06-11; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Prospective Cohort Study of Synovial Biomarkers in the Diagnosis and Prediction of Periprosthetic Joint Infection
Keywords: Prospective cohort study; synovial biomarkers; diagnosis; prediction; periprosthetic joint infection
MeSH Terms: conditions — Disease | interventions — Arthrocentesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Synovial fluid aspirating from patients' joint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infection group: Joint puncture to extract joint fluid
  Interventions: Device: Joint aspiration
- None infection group: Joint puncture to extract joint fluid
  Interventions: Device: Joint aspiration

INTERVENTIONS:
Device: Joint aspiration — Joint puncture to extract joint fluid.

SUMMARY:
Prosthetic Joint Infection (PJI) is one of the severe complications following arthroplasty. With the global aging population, the number of patients undergoing primary joint replacement surgeries is increasing, leading to a rise in PJI cases. Although the incidence of PJI is generally low, the impact on patients can be catastrophic. Once an infection occurs, it is further complicated by the rising global antibiotic resistance, imposing a significant economic burden on patients. Therefore, improving the diagnostic rate of PJI is crucial. Currently, various infection markers are used in the diagnosis of PJI. However, there is still a lack of highly sensitive and specific markers to effectively diagnose PJI, necessitating the exploration of new infection markers. This study aims to investigate novel infection markers for the diagnosis of PJI, providing evidence for its diagnosis and subsequent treatment. In this research, we will prospectively collect data from patients undergoing primary joint replacement and those developing PJI from June 2024 to December 2026. These patients will be categorized into non-infection and infection groups. By collecting and analyzing general patient data, surgery-related information, and infection-related indicators from preoperative joint fluid and blood samples, we aim to further evaluate the predictive value of these infection markers for PJI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender is not limited;
2. The experimental group met the diagnostic criteria of chronic periprosthesis infection after joint replacement according to the 2018 Musculoskeletal Infection Association; The control group was eligible for primary replacement patients who excluded periprosthesis infection.
3. Voluntary and signed informed consent.

Exclusion Criteria:

1. Patients with immune-related arthritis such as rheumatoid and rheumatism were excluded;
2. Radiotherapy and chemotherapy are required due to neoplastic diseases;
3. Receiving systemic glucocorticoid therapy (prednisone > 10mg/ day or equivalent hormone medication);
4. Severe immunodeficiency diseases (such as stage 3 HIV, sickle cell anemia, splenectomy, etc.);
5. Have a history of drug abuse;
6. Use immunosuppressive drugs to treat bone marrow or other transplants;
7. Pregnant, parturient and lactating women;
8. Participating in other clinical trials;
9. Researchers consider other reasons not appropriate for clinical trial participants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with periprosthesis infection or non-periprosthesis infection
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Joint fluid target protein detection | One day before surgery or one day after surgery
  To detect new target proteins by elisa test.

SECONDARY OUTCOMES:
X-ray | One day before surgery and two years after surgery
  X-ray of surgery site.
Erythrocyte sedimentation rate (ESR) | One day before sugery and two year after surgery
  It measures the rate at which red blood cells settle to the bottom of a test tube within one hour.
  Normal ranges:
  Male: 0 to 15 millimeters per hour (mm/hr) Female: 0 to 20 millimeters per hour (mm/hr)
C-reactive protein (CRP) | One day before sugery and two year after surgery
  C-reactive protein (CRP) is a protein produced by the liver that significantly increases in response to inflammation or infection. Normal range for CRP is less than 10 milligrams per liter (mg/L).
Synovial fluid white blood cell count (SF-WBC) | One day before surgery and one day after surgery
  Synovial fluid white blood cell count (SF-WBC)
Synovial fluid polymorphonuclear cells (SF-PMN) | One day before surgery and one day after surgery
  Polymorphonuclear neutrophil percentage in synovial fluid refers to the proportion or percentage of polymorphonuclear neutrophils (PMN) present in the synovial fluid. This measurement is important in the assessment of joint health and inflammation, particularly in conditions such as arthritis and infections affecting the joints. Normal range: Less than 80%.
Doppler lower extremity vascular color ultrasound | One day before surgery and three day after surgery
  Doppler lower extremity vascular color ultrasound to evaluate the deep vein thrombus development
American Knee Society Score (AKS score) | One day before surgery, two years after surgery
  American Knee Society Score is used to evaluate the outcomes of knee replacement surgery. This scoring system consists of two main components: the knee score and the function score.
  Knee Score: This primarily assesses the condition of the knee joint itself, including pain, stability, and range of motion. The higher of the score, the better of the functional result.
The Hip Harris Score (HHS) | One day before surgery, two years after surgery
  The Harris Hip Score (HHS) is a widely used clinical tool for assessing the outcomes of hip surgeries, particularly hip replacements. Developed by Dr. William Harris in 1969, it evaluates various aspects of hip function and pain to provide an overall score that reflects the patient's condition. The higher the score, the better the result is.
Alanine Aminotransferase (ALT) | One day before surgery and one day after surgery
  An enzyme found in the liver that helps convert proteins into energy. Elevated levels indicate liver damage. Normal range: 10 to 40 units per liter (U/L)
Aspartate Aminotransferase (AST) | One day before surgery and one day after surgery
  An enzyme found in the liver and other tissues. High levels can indicate liver damage but are less specific than ALT. Normal range: 10 to 40 units per liter (U/L)
Serum Creatinine | One day before surgery and one day after surgery
  Measures the level of creatinine in the blood. Elevated levels can indicate impaired kidney function. Normal range: 62 to 115 micromoles per liter (µmol/L).
Blood Urea Nitrogen （BUN） | One day before surgery and one day after surgery
  Measures the amount of nitrogen in the blood that comes from urea. Elevated BUN levels can indicate impaired kidney function. Normal range: 2.5 to 7.1 millimoles per liter (mmol/L).

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be acquired from corresponding author by reasonable reason.
Supporting Information: Study Protocol
Time Frame: After our paper published.